CLINICAL TRIAL: NCT05179798
Title: The Study of Recommendation System DiaCompanion With Personalized Dietary Recommendations for Women With Gestational Diabetes Mellitus (DiaCompanion I)
Brief Title: The Study of Recommendation System DiaCompanion for Women With Gestational Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Responsible Party: Principal Investigator, Polina Popova, Head of the research laboratory of methabolic disorders and microbiota, Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DiaCompanion I
Record Dates: First submitted 2021-10-30; First posted 2022-01-05 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Gestational Diabetes Mellitus (GDM)
Keywords: gestational diabetes mellitus; glycemic targets; mHealth; personalized medicine; recommendation system; personalized nutrition; postprandial glycemic response
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile app (Experimental): Lifestyle modification, insulin therapy if needed, utilization of a mobile app with personalized recommendations.
  Interventions: Device: mobile app
- Standard of care (No Intervention): Lifestyle modification, insulin therapy if needed; conventional care without a mobile app.

INTERVENTIONS:
Device: mobile app — Lifestyle modification, insulin therapy if needed, utilization of a mobile app with personalized recommendations.
  Other Names: recommendation system
  Arms: Mobile app

SUMMARY:
This is a randomized controlled trial of a recommendation system implementation in the treatment of women with gestational diabetes mellitus (GDM). The trial assesses the aspects of system effects on maternal glucose control, the fetus and pregnancy outcomes. This study is an interventional, randomized controlled trial, open-labeled.

DETAILED DESCRIPTION:
The study aims to clarify the effect of using DiaCompanion I (a mobile-based personalized recommendations system) on glycemic levels and pregnancy outcomes in women with GDM. Women with GDM are randomized to 2 treatment groups (utilizing and not utilizing the developed mobile-based system with data-driven personal recommendations focused primarily on postprandial glycemic response prediction). Data on glycemic levels during the study and consumption of major macro- and micronutrients will be collected using the mobile app with electronic report forms. The app provides women in the intervention group with the resulting data-driven prognosis of a 1-hour postprandial glucose level every time they input their meal data. The app also provides participants of the intervention group with a set of reminders and recommendations on the diet and lifestyle.

Apart from the assessment of the outcomes described below, biobanking of serum, plasma; cord fluid, HUVECs, faeces, and meconium will be performed. The samples may be used for further analyses in ancillary studies, which could be beneficial for GDM care based on evolution in scientific knowledge.

This biological collection is optional [Time Frame: within 15 years after the end of the study]:

* The blood samples will be collected at the same time as the sample routinely collected
* Maternal faeces will be collected within 5 days after inclusion and at gestational weeks 35-36
* Cord fluid will be collected
* HUVECs will be isolated from the cord after delivery
* Meconium will be collected within 24 hours after birth.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with GDM according to IADPSG (International Association of the Diabetes and Pregnancy Study Groups) criteria, i.e. fasting plasma glucose between 5.1 mmol/L and 6.9 mmol/L after the 6th week of gestation and/or 1-hour plasma glucose value after 75 g oral glucose tolerance test (OGTT) ≥ 10.0 mmol/L and/or 2-hour plasma glucose value between 8.5 mmol/L and 11.0 mmol/L at the 24-31st week of gestation
* Age >18 years
* Gestational age >= 12 and < 32 weeks
* No more than 4 weeks after confirmation of GDM diagnosis
* Singleton pregnancy
* The ability to navigate an app
* Provided informed consent

Exclusion Criteria:

* Preexisting diabetes of any type before the current pregnancy
* Need for insulin therapy at the time of screening
* Heart failure
* Chronic kidney disease
* History of bariatric surgery
* Use of long-term systemic corticosteroids
* Impaired mobility
* Known fetal malformations
* Concomitant participation in other clinical trials

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 216 (Estimated)
Dates: Start 2022-01-12 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of postprandial capillary glucose values above target (>7.0 mmol/L) | from randomization up to delivery
  The women will be asked to perform 6 measures a day. Capillary glucose values will be retrieved from the glucose meter, and if not available, from the woman's diary.

SECONDARY OUTCOMES:
Rate of patients requiring insulin therapy during pregnancy | At any time during pregnancy up to delivery
  * Rate of patients requiring insulin therapy (either basal or prandial)
  * Rate of patients requiring prandial insulin therapy
Capillary glucose values | within 2 weeks after randomization, at gestational weeks 35-37 and in the period from randomization up to delivery
  The women will be asked to perform 6 measures a day. Capillary glucose values will be retrieved from the glucose meter and from the woman's diary.
  * Capillary fasting glucose values, mmol/L
  * Capillary pre-prandial glucose values, mmol/L
  * Capillary postprandial glucose values, mmol/L
Proportion of women with glucose values within target | within 2 weeks after randomization, at gestational weeks 35-37 and in the period from randomization up to delivery
  * The proportion of women with fasting glucose values within the target
  * The proportion of women with postprandial glucose values within the target
Mean incremental area under the blood glucose curve 2 hours after meals (iAUC120) according to continuous glucose monitoring (time period: 7 days) | 1-2 weeks after randomization and 35-37th gestational week
Hypoglycemia | from randomization to delivery
  * Severe hypoglycemia: requiring assistance of another person to actively correct the level of glycemia and neurological symptoms
  * Documented symptomatic hypoglycemia: event during which typical symptoms of hypoglycemia are accompanied by a measured capillary glucose concentration <3.9 mmol/L
  * Asymptomatic hypoglycemia: event not accompanied by typical symptoms of hypoglycemia but with a measured capillary glucose concentration <3.3 mmol/L
The level of HbA1c, % | at gestational weeks 35-37
  Maternal metabolic parameter: The level of HbA1c, %
Fasting insulin, mIU/mL | at gestational weeks 35-37
  Maternal metabolic parameter: Fasting insulin, mIU/mL
Fasting glucose, mmol/L | at gestational weeks 35-37
  Maternal metabolic parameter: Fasting glucose, mmol/L
HOMA-IR index | at gestational weeks 35-37
  Maternal metabolic parameter: HOMA-IR index
Serum triglyceride levels, mmol/L | at gestational weeks 35-37
  Maternal metabolic parameter: Serum triglyceride levels, mmol/L
Gestational weight change | by the time of delivery
  * Gestational weight change during pregnancy, kg
  * Gestational weight change between inclusion and delivery, kg
Large (>90th percentile) for gestational age infant | At delivery
  Neonatal outcome: Large (>90th percentile) for gestational age infant
Small for gestational age (< 10th percentile) infant | At delivery
  Neonatal outcome: Small for gestational age (< 10th percentile) infant
Birth weight, kg | At delivery
  Neonatal outcome: Birth weight, kg
Birth weight ≥ 4000 g; ≥ 4500 g | At delivery
  Neonatal outcome: Birth weight ≥ 4000 g; ≥ 4500 g (yes/no)
Neonatal hypoglycemia | At delivery
  Neonatal outcome: Neonatal hypoglycemia (yes/no)
Shoulder dystocia | At delivery
  Neonatal outcome: Shoulder dystocia (yes/no)
Birth injury, any of the following: plexus injury, clavicle, humeral, or skull fracture | At delivery
  Neonatal outcome: Birth injury, any of the following: plexus injury, clavicle, humeral, or skull fracture (yes/no)
Preterm delivery | At delivery
  Neonatal outcome: Preterm delivery (yes/no)
Apgar score at 1 and 5 minutes from birth | At delivery
  Neonatal outcome: Apgar score at 1 and 5 minutes from birth
Low Apgar score: 5-min Apgar score < 7 | At delivery
  Neonatal outcome: Low Apgar score: 5-min Apgar score < 7
Jaundice requiring phototherapy | At delivery
  Neonatal outcome: Jaundice requiring phototherapy (yes/no)
Neonatal respiratory distress syndrome | At delivery
  Neonatal outcome: Neonatal respiratory distress syndrome (yes/no)
Admission to neonatal intensive care unit during the three days following birth | At delivery
  Neonatal outcome: Admission to neonatal intensive care unit during the three days following birth (yes/no)
Umbilical cord blood C-peptide, ng/mL | At delivery
  Neonatal outcome: Umbilical cord blood C-peptide, ng/mL
Cesarean delivery rate | At any time during pregnancy up to delivery
  Maternal outcome: Cesarean delivery rate
Induction of labor rate | At any time during pregnancy up to delivery
  Maternal outcome: Induction of labor rate
Need for operative vaginal delivery rate | At any time during pregnancy up to delivery
  Maternal outcome: Need for operative vaginal delivery rate (forceps or vacuum-assisted vaginal delivery)
Preeclampsia | At any time during pregnancy up to delivery
  Maternal outcome: Preeclampsia (blood pressure ≥ 140/90 mmHg on two measurements four hours apart and proteinuria of at least 300 mg/24 hours or 3+ or more on dipstick testing or proteinuria/creatinuria >30 in a random urine sample)
Pregnancy-induced hypertension in women with no known hypertension before pregnancy | At any time during pregnancy up to delivery
  Maternal outcome: Pregnancy-induced hypertension in women with no known hypertension before pregnancy, blood pressure ≥ 140/90 mmHg on two measurements four hours apart without proteinuria and having needed to begin anti-hypertensive therapy
The number of in-patient visits to endocrinologists | from randomization to delivery
Results of oral glucose tolerance test | 3 months after delivery
  The test will be performed by the women 3 months postpartum
Acceptance/satisfaction of 2 strategies: score | at gestational weeks 35-36
  Evaluation of the patient's satisfaction about their treatment for GDM with a scale: give a score of 0 to 100: 0 not satisfied; 100 totally satisfied
Patient satisfaction evaluated through a questionnaire | at gestational weeks 35-36
  10-question questionnaire with multiple-choice questions, questions with numeric answers on the scale from 0 (fully unsatisfied) to 10 (fully satisfied) and open-ended questions

CONTACTS AND LOCATIONS:
Locations (1):
- Almazov National Medical Research Centre, Saint Petersburg, Russia

REFERENCES:
- [Background] Pustozerov E, Tkachuk A, Vasukova E, Dronova A, Shilova E, Anopova A, Piven F, Pervunina T, Vasilieva E, Grineva E, Popova P. The Role of Glycemic Index and Glycemic Load in the Development of Real-Time Postprandial Glycemic Response Prediction Models for Patients With Gestational Diabetes. Nutrients. 2020 Jan 23;12(2):302. doi: 10.3390/nu12020302. PMID 31979294
- [Background] Pustozerov E.A., Tkachuck A.S., Vasukova E.A., Anopova A.D., Kokina M.A., Gorelova I.V., Pervunina T.M., Grineva E.N., Popova P.V. Machine Learning Approach for Postprandial Blood Glucose Prediction in Gestational Diabetes Mellitus. IEEE Access, vol. 8, pp. 219308-219321, 2020, doi: 10.1109/ACCESS.2020.3042483.
- [Background] Pustozerov E, Popova P, Tkachuk A, Bolotko Y, Yuldashev Z, Grineva E. Development and Evaluation of a Mobile Personalized Blood Glucose Prediction System for Patients With Gestational Diabetes Mellitus. JMIR Mhealth Uhealth. 2018 Jan 9;6(1):e6. doi: 10.2196/mhealth.9236. PMID 29317385
- [Derived] Popova P, Anopova A, Vasukova E, Isakov A, Eriskovskaya A, Degilevich A, Pustozerov E, Tkachuk A, Pashkova K, Krasnova N, Kokina M, Nemykina I, Pervunina T, Li O, Grineva E, Shlyakhto E. Trial protocol for the study of recommendation system DiaCompanion with personalized dietary recommendations for women with gestational diabetes mellitus (DiaCompanion I). Front Endocrinol (Lausanne). 2023 Jun 7;14:1168688. doi: 10.3389/fendo.2023.1168688. eCollection 2023. PMID 37361536